CLINICAL TRIAL: NCT03384251
Title: Assessing an Educational Intervention Program on Knowledge, Attitude and Behaviour Towards Pregnancy Prevention Based on Health Belief Model Amongst Adolescent Girls in Northern Ghana: A Clustered Randomized Trial
Brief Title: Assessing an Educational Intervention Program on Knowledge, Attitude and Behaviour Towards Pregnancy Prevention Based on Health Belief Model Amongst Adolescent Girls in Northern Ghana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ibrahim Yakubu, Principal Investigator, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IR.TUMS.SPH.REC.1396.4089; GHS-ERC:020-03-18 (Other: Ghana Health Service Ethics Review Committee)
Record Dates: First submitted 2017-12-16; First posted 2017-12-27 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-09

CONDITIONS: Adolescent Behavior
Keywords: Adolescent pregnancy; Teenage pregnancy; Prevention; Ghana
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: A multi-stage sampling method shall be conducted. A random sampling of six (6) out 12 mixed Senior High Schools in Tamale Metropolis-Northern Ghana would be selected. We shall randomly allocate three (3) schools as the intervention and the other three (3) as control groups respectively. In each school, one class shall be selected at random from each grade in both intervention and control groups.
Masking Description: Participants are not required to write their names on the questionnaires. therefore responses provided are anonymous
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): This group shall be given a comprehensive sex education in approximately six sessions.
  Interventions: Behavioral: comprehensive sex education
- Control group (No Intervention): This group will not be given any form of education.

INTERVENTIONS:
Behavioral: comprehensive sex education — A comprehensive sex education program to be delivered in approximately six (6) sessions comprising of an introductory lesson on susceptibility and severity of teenage pregnancy, personal and community values, female reproductive system, contraception and decision-making skills.
  Arms: Intervention group

SUMMARY:
The study is designed to assess the impact of an educational intervention program on the knowledge, attitude and behaviour towards pregnancy prevention based on Health Belief Model amongst adolescent girls in Northern Ghana. It is a randomised clustered controlled trial to be conducted on Senior High School students in Northern Ghana The study hypothesises that knowledge, attitude and behaviour of adolescents towards pregnancy prevention will differ between the groups.

DETAILED DESCRIPTION:
Adolescent pregnancy is a global problem because of its health, social, economic and political repercussions on the globe. According to WHO about 16 million girls aged 15 to 19 and some 1 million girls under 15years give birth every year, mostly in low and middle-income countries. Babies born to adolescent mothers face a substantially higher risk of dying than those born to women aged 20 to 24. Pregnant adolescents also develop psychological problems from social stigma, suffering physical and domestic violence in her attempt to meeting the demands of pregnancy and childbearing. Children born to adolescents are at risk of malnutrition, low mental and physical development, inappropriate social connection with parents and poor education.

The factors associated with adolescent pregnancies include early marriages, poor social and economic support. Curiosity and peer pressure, lack of sexuality education, poor reproductive health services and poor attitude of health workers to providing contraceptive services for adolescents amongst others.

Ghana developed a number of policies to improve adolescent development through the provision of youth focus friendly health services in the country. However, adolescent pregnancy has not declined as expected.

The Health Belief Model is one of the appropriate health promotion models designed to predict preventive health behaviours, and it has enhanced preventive health behaviours in breast cancer screening and prevention of risky sexual behaviours in adolescents as well as prevention of iron deficiency anaemia. Schools are the best site for providing health education and promotion interventions because students spend most of the time in school and health promoters have the opportunity of reaching a large number of participants. Students of Senior High Schools in Ghana are adolescents and most of them are sexually active and has little knowledge about sex education and use of contraceptives. Therefore, providing comprehensive sex education to adolescents in schools will increase their knowledge; enhance their attitude and behavior towards pregnancy prevention.

This study, therefore, is intended to assess the impact of an educational intervention program on the knowledge, attitude and behavior towards pregnancy prevention based on Health Belief Model amongst adolescent girls in Northern Ghana.

The main objective is to assess the impact of an educational intervention program on knowledge, attitude and behavior towards pregnancy prevention based on Health Belief Model amongst adolescent girls in Northern Ghana.

Study design: The study shall be an interventional research using Clustered Randomized Controlled Trial to assess the impact of an educational program on the knowledge, attitude and behavior of adolescents towards teenage pregnancy using a researcher-structured questionnaire based on the Health Belief Model and a validated psychometric "Teen Attitude Pregnancy Scale" Intervention: A comprehensive sex education program shall be delivered in approximately six (6) sessions comprising of an introductory lesson on susceptibility and severity of teenage pregnancy, personal and community values, female reproductive system, contraceptives and decision-making. A qualified midwife shall conduct the health education program. Teaching and learning materials shall include flip charts, contraceptives, short videos, role-play scenarios among others. A practical demonstration, group discussion, lectures, role-play and interactive learning methods shall be employed. Attitudinal and behavioural intervention strategies shall be adopted for the study based on the Taxonomy of Behavior Change Techniques for interventions

ELIGIBILITY:
Inclusion Criteria:

* Only unmarried adolescent female high school students shall be included in the study.

Exclusion Criteria:

* Girls who do not want to participate and those who do not fall within the adolescent age group as well as married adolescents shall be excluded

Ages: 13 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Only female adolescents are to participate in this study
Enrollment: 363 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Health Belief Model constructs | 3 months and 6 months
  A questionnaire designed by the researchers based on the HBM six constructs shall be used to assess adolescents perception towards pregnancy prevention. A total of 58 items were used.
  The items specifically assess adolescents' opinion on their chances of getting pregnant; adolescents' opinion on the seriousness of adolescent pregnancy and the consequences of getting pregnant; adolescents' opinion on the importance delaying pregnancy, adolescents' opinion on the barriers of delaying pregnancy; and adolescents' confidence on their ability to delay pregnancy.
  The degree with which participants perceived each of these items were recorded using a five-point Likert's scale ranging from "strongly disagree for a lower score to strongly agree for a higher score". Each domain has the same minimum score of zero (0) and a maximum score of 40. All the scores for the HBM domain variables shall be expressed in percentages for analysis.

SECONDARY OUTCOMES:
Abstinence from sexual intercourse | 3 months and 6 months
  Two (2) questions shall be used to assess abstinence practice. One question will assess participants' intention to abstain from sexual intercourse.
  Abstinence practice is a binary variable where a score of one (1) will be labelled "yes" and Zero (0) labelled "no". The question on intention is on a three-scale item; 1=definitely will, 2=not sure and 3=definitely won't. A score of one denotes low abstinence intention and a score of three denotes high abstinence intention. The intention scores shall be expressed in percentages for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Yakubu, Principal Investigator — Tehran University of Medical Sciences
Locations (2):
- Ghana (2):
  - Kalpohin Senior High School, Tamale, Northern Region
  - Vittin Senoir High School, Tamale, Northern Region

IPD SHARING:
Plan to Share IPD: Yes
The data may be shared on request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after the study
Access Criteria: If data is requested especially by journals it would be sent by email.

REFERENCES:
- [Background] Ganchimeg T, Ota E, Morisaki N, Laopaiboon M, Lumbiganon P, Zhang J, Yamdamsuren B, Temmerman M, Say L, Tuncalp O, Vogel JP, Souza JP, Mori R; WHO Multicountry Survey on Maternal Newborn Health Research Network. Pregnancy and childbirth outcomes among adolescent mothers: a World Health Organization multicountry study. BJOG. 2014 Mar;121(Suppl 1):40-8. doi: 10.1111/1471-0528.12630. PMID 24641534
- [Background] Aransiola JO, Asa S, Obinjuwa P, Olarewaju O, Ojo OO, Fatusi AO. Teachers' perspectives on sexual and reproductive health interventions for in-school adolescents in Nigeria. Afr J Reprod Health. 2013 Dec;17(4):84-92. PMID 24558785
- [Background] Atuyambe L, Mirembe F, Johansson A, Kirumira EK, Faxelid E. Experiences of pregnant adolescents--voices from Wakiso district, Uganda. Afr Health Sci. 2005 Dec;5(4):304-9. doi: 10.5555/afhs.2005.5.4.304. PMID 16615840
- [Background] Ahorlu CK, Pfeiffer C, Obrist B. Socio-cultural and economic factors influencing adolescents' resilience against the threat of teenage pregnancy: a cross-sectional survey in Accra, Ghana. Reprod Health. 2015 Dec 23;12:117. doi: 10.1186/s12978-015-0113-9. PMID 26700638
- [Background] Krugu JK, Mevissen FE, Prinsen A, Ruiter RA. Who's that girl? A qualitative analysis of adolescent girls' views on factors associated with teenage pregnancies in Bolgatanga, Ghana. Reprod Health. 2016 Apr 14;13:39. doi: 10.1186/s12978-016-0161-9. PMID 27080996
- [Background] Abdul-Rahman L, Marrone G, Johansson A. Trends in contraceptive use among female adolescents in Ghana. Afr J Reprod Health. 2011 Jun;15(2):45-55. PMID 22590892
- [Background] Adinma JI, Agbai AO, Okeke AO, Okaro JM. Contraception in teenage Nigerian school girls. Adv Contracept. 1999;15(4):283-91. doi: 10.1023/a:1006732222373. PMID 11145370
- [Background] Somers CL, Johnson SA, Sawilowsky SS. A measure for evaluating the effectiveness of teen pregnancy prevention programs. Psychology in the Schools. 2002;39(3):337-42.
- [Background] Yidana A, Ziblim S-D, Azongo TB, Abass YI. Socio-Cultural Determinants of Contraceptives Use Among Adolescents in Northern Ghana. Public Health Research. 2015;5(4):83-9.
- [Result] World Health Organization: Adolescent pregnancy Fact sheet [Internet]. World Health Organization. 2014 [cited September 2014]. Available from: http://www.who.int/mediacentre/factsheets/fs364/en/.
- [Derived] Yakubu I, Garmaroudi G, Sadeghi R, Tol A, Yekaninejad MS, Yidana A. Assessing the impact of an educational intervention program on sexual abstinence based on the health belief model amongst adolescent girls in Northern Ghana, a cluster randomised control trial. Reprod Health. 2019 Aug 15;16(1):124. doi: 10.1186/s12978-019-0784-8. PMID 31416450